CLINICAL TRIAL: NCT04423939
Title: ACT to Reduce Morbidity and Mortality in Hematopoietic Stem Cell Transplant (HCT) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00105683
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic Steam Cell Transplantation (HCT)
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hematopoietic Stem Cell Transplantation (HCT) Patients (Experimental): 20 HCT patients at Duke
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Caregivers (Experimental): 20 HCT patients caregivers at Duke
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — The ACT sessions will be tailored to the clinical challenges of HCT. Sessions are with a mental health professional and are 45-60 minutes in duration and include both the participant and caregiver.

SUMMARY:
This is a research study to develop and test a novel protocol to reduce physical and psychological vulnerabilities that contribute to treatment intolerance and treatment-related morbidity and mortality among hematopoietic stem cell transplant (HCT) patients. When the participant enrolls in this study, they will be asked to participate in acceptance and commitment therapy (ACT) as well as complete in-person physical function tests and a cognitive test. They will also receive training on how to use iOS devices (e.g. iPad, iPhone) and activity trackers (e.g. Apple Watch), which will be provided to them during the duration of study participation. The study team will ask you to complete multiple surveys about emotional and cognitive function, diet and social support, and ask the participant to provide feedback about the treatment (e.g., what they liked or did not like). The study team will also ask the participant to provide stool samples for analysis of the bacteria in intestines, skin surface swabs for analysis of the bacteria on skin and blood samples for analysis of biomarkers and metabolites. Biomarkers and metabolites are molecular and cellular parts that deal with genetic makeup, like DNA, RNA, protein, and/or other naturally occurring substances that may be associated with transplant outcomes. Participants can expect to be enrolled in this study for 3 years.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Over the age of 18
* Undergoing allogeneic HCT for any cancer or noncancer illness
* English speaking
* Has a caregiver willing to participate

Caregiver:

* Over the age of 18
* English speaking

Exclusion Criteria:

* Under the age of 18
* Non-English speaking
* Has a caregiver unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2025-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sung, MD, Principal Investigator — Duke University
Locations (1):
- Lauren Hill, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Duke Adult Bone Marrow Transplant program between August 2020 and September 2022. The first subject was consented on October 14, 2020 and the last subject was consented on June 7, 2022.
Pre-assignment Details: Five subjects consented to the study but were excluded before starting intervention. One patient's caregiver declined to participate and lack of caregiver participation is an exclusion criteria for this study. One patient was no longer scheduled to receive an allogeneic transplant and they and their caregiver were excluded. One patient relapsed and was no longer getting a transplant and they and their caregiver were excluded.
Groups:
- Hematopoietic Stem Cell Transplantation (HCT) Patients: HCT patients at Duke
  Acceptance and Commitment Therapy (ACT): The ACT sessions will be tailored to the clinical challenges of HCT. Sessions are with a mental health professional and are 45-60 minutes in duration and include both the participant and caregiver.
- Caregivers: HCT patient caregivers at Duke
  Acceptance and Commitment Therapy (ACT): The ACT sessions will be tailored to the clinical challenges of HCT. Sessions are with a mental health professional and are 45-60 minutes in duration and include both the participant and caregiver.
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation (HCT) Patients | Caregivers
Started | 14 | 14
Completed | 0 | 0
Not Completed | 14 | 14
Not completed — Still on study (but completed primary endpoint) | 8 | 8
Not completed — Death | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Caregiver to patient who died | 0 | 3
Not completed — Caregiver to patient who withdrew | 0 | 3

BASELINE CHARACTERISTICS:
Population: 14 patients and their caregivers were included in the analysis for this study.
Groups:
- Hematopoietic Stem Cell Transplantation (HCT) Patients: 14 HCT patients at Duke
  Acceptance and Commitment Therapy (ACT): The ACT sessions will be tailored to the clinical challenges of HCT. Sessions are with a mental health professional and are 45-60 minutes in duration and include both the patient and caregiver.
- Caregivers: 14 HCT patients' caregivers at Duke
  Acceptance and Commitment Therapy (ACT): The ACT sessions will be tailored to the clinical challenges of HCT. Sessions are with a mental health professional and are 45-60 minutes in duration and include both the patient and caregiver.
- Total: Total of all reporting groups
Arm/Group | Hematopoietic Stem Cell Transplantation (HCT) Patients | Caregivers | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (14.6) | 58.1 (11.9) | 55.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Diagnosis [Count of Participants; unit: Participants] — Population: Caregivers are not included in the diagnosis category
  Participants
    number analyzed (Participants) | 14 | 0 | 14
    Acute myeloid leukemia | 6 |  | 6
    Myeloproliferative neoplasm | 3 |  | 3
    Myelodysplastic syndrome | 2 |  | 2
    Diffuse large B cell lymphoma | 1 |  | 1
    Acute lymphoblastic leukemia | 1 |  | 1
    Chronic myeloid leukemia | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Function, as Measured by 6 Minute Walk Test (6MWT)
Description: The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Time Frame: Baseline (~30 days before HCT), Signoff (~10 days before HCT), Day 90 post-HCT
Measure: Mean (95% Confidence Interval); unit: meters
Groups:
- Hematopoietic Stem Cell Transplantation (HCT) Patients: 14 HCT patients at Duke
  Acceptance and Commitment Therapy (ACT): The ACT sessions will be tailored to the clinical challenges of HCT. Sessions are with a mental health professional and are 45-60 minutes in duration and include both the participant and caregiver.
Arm/Group | Hematopoietic Stem Cell Transplantation (HCT) Patients
Number analyzed (Participants) | 14
meters
  Baseline (~30 days before HCT) | 449 [421 to 477]
  Sign off (~10 days before HCT) | 468 [439 to 496]
  Day 90 | 478 [447 to 509]

2. Primary Outcome: Hospital Length of Stay, as Measured by Medical Record Review
Description: Hospital length of stay in days
Time Frame: Up to Day 90
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Hematopoietic Stem Cell Transplantation (HCT) Patients
Number analyzed (Participants) | 14
days | 31.4 (27.6)

3. Other Pre Specified Outcome: Change in Shannon Diversity, as Measured by Stool Samples
Description: Stool samples assessed by 16s rRNA sequencing
Time Frame: Baseline, Day 90
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Shannon Diversity, as Measured by Stool Samples
Description: Stool samples assessed by 16s rRNA sequencing
Time Frame: Baseline, D0, D7, D14, D21, Day 30, Day 60, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Hospital Length of Stay, as Measured by Medical Record Review
Description: Hospital length of stay in days
Time Frame: Up to 3 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Physical Function, as Measured by 6 Minute Walk Test
Description: The baseline for each patient is made through an algorithm that factors the patients age and gender. The patient's score is compared to what a person that is the patient's same age and gender would get. This comparison is then used as a tool to assess aerobic capacity or endurance.
Time Frame: Baseline, Day 30, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Clinical Outcomes, as Assessed by Adverse Events Reporting
Description: Post-HCT clinical outcomes (i.e. GVHD)
Time Frame: Continuous from baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Acceptability of the Intervention, as Assessed by Exit Interviews
Description: Exit interviews to assess patients' opinion on the ACT program
Time Frame: Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Acceptability of the Intervention, as Assessed by the Acceptability Survey
Description: 6-item survey to assess patients' opinion on the ACT program
Time Frame: Baseline, at each ACT session time point
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Flow Cytometry, as Measured by Blood Samples
Description: Whole blood samples, will be analyzed and monitored for outcomes such as immune cell differentiation, immune response and development of GVHD. Flow cytometry will be performed.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in Metabolomics, as Measured by Blood Samples
Description: Approximately 1ml of plasma from the EDTA tube will be used for metabolomics analysis.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Changes in Biomarkers, as Measured by Blood Samples
Description: Assays evaluating angiogenic, stromal, and inflammatory markers and markers of aging (the Pepper Panel) are used to assess inflammation and frailty.
Time Frame: Baseline, Day 14, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Microbiome Diversity, as Measured by Skin Swabs
Description: Skin swab samples batch sequenced and microbiome analyzed
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Symptom Severity, as Measured by PRO-CTCAE Core Symptom Assessment
Description: Assessing changes in severity of core symptoms that are typically associated with HCT
Time Frame: Day 0, Year 1
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Overall Well-being, as Measured by PROMIS Sleep Assessment
Description: The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Overall Well-being, as Measured by PROMIS Global Health Assessment
Description: as for outcome 15
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Caregiver Quality of Life, as Measured by Self-Efficacy and Preparedness for Caregivers Assessment
Description: 9-item questionnaire to assess preparedness for caregiving
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in Quality of Life, as Measured by Lorig Self-Efficacy Assessment
Description: The Self-Efficacy to Manage Chronic Disease Scale is made up of 6-items on a visual analog scale, ranging from 1 (not at all confident) to 10 (totally confident).
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Quality of Life, as Measured by EQ-5D-5L Assessment
Description: The 5D represents 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Five levels of severity are measured, as indicated by the "5L," ranging from "no problems" to "extreme problems." All scores are converted into a summary index.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Caregiver Quality of Life, as Measured by FACT-GP Assessment
Description: 21 item assessment scored on a 5-point Likert scale
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change in Quality of Life, as Measured by FACT-BMT Assessment
Description: 50 item assessment. Higher total and domain scores indicate greater quality of life.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Change in Overall Well-being, as Measured by OARS IADLs Assessment
Description: OARS IADL is a 7 item assessment that asks what level of assistance is needed to do 7 different activities of daily living
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Change in Overall Well-being, as Measured by Fried Frailty Assessment
Description: The scores of all of the sections are added and if the patient has a score greater or equal to three this assessment deems that the patients is frail. If the patient has a score between 1-2 the patient is deemed pre-frail.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Change in Financial Status, as Measured by Financial Assessment
Description: 22-item questionnaire to assess how a patient's care as affected their finances
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Change in Caregiver Socioeconomic Status, as Measured by SES Assessment
Description: Questionnaire to assess caregiver socioeconomic status
Time Frame: Baseline, D180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Change in Financial Status, as Measured by COST-FACIT Assessment
Description: COST-FACIT is an 11-item questionnaire that assesses a patient's financial toxicity
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Change in Social Well-being, as Measured by CMS Social Determinants of Health (SDOH) Assessment
Description: CMS SDOH is a 10 item survey that assesses 5 domains of social needs
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Change in Nutrition, as Measured by ASA-24 Assessment
Description: ASA-24 is a self-administered 24-hour diet recall
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Change in Nutrition, as Measured by PG-SGA/Clinician SGA Assessment
Description: Scores for each section can range from 0-4 depending on severity and nutritional impact. The sum of all scores provides the Total PG-SGA score, which can be used to indicate the need for intervention (Bauer et al., 2002)
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Change in Nutrition, as Measured by Perioperative Nutrition Screen (PONS)
Description: PONS analyzes BMI, weight loss, and food intake to screen for preoperative nutrition risk
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Change in Nutrition, as Measured by Body Mass Index (BMI)
Description: BMI can be associated with a patient's nutritional health
Time Frame: Continuous from baseline
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Change in Nutrition, as Measured by Albumin Values
Description: Albumin levels can be associated with a patient's nutritional health
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Change in Mental Health, as Measured by Brief COPE Assessment
Description: Scores are presented for three overarching coping styles as average scores (sum of item scores divided by number of items), indicating the degree to which the respondent has been engaging in that coping style.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Change in Mental Health, as Measured by HHI-12 Assessment
Description: The HHI-12 is an adapted 12 question version of the Hearth Hope Scale that assesses a patient's sense of hope
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Change in Mental Health, as Measured by PROMIS Social Isolation Assessment
Description: as for outcome 15
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Change in Mental Health, as Measured by PROMIS Emotional Support Assessment
Description: as for outcome 15
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Change in Mental Health, as Measured by PROMIS Anxiety Assessment
Description: as for outcome 15
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Change in Mental Health, as Measured by PROMIS Depression Assessment
Description: as for outcome 15
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Change in Mental Health, as Measured by PC-PTSD/PCL-5 Assessment
Description: PC-PTSD is a 5 item screen to identify patients with probable PTSD. If the patient screens positive, they then take the PCL-5. The PCL-5 is a 20 item screen to assess symptoms of PTSD.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Target Engagement (Process of Change), as Assessed by Valuing Questionnaire (VQ)
Description: The VQ is a 10-item self-report questionnaire that assesses how closely a person is living in align with their values over the last week. Progress (range = 0 to 30) is defined as enactment and perseverance in living consistently with one's values; higher scores represent a closer alignment between one's internal values and one's actions. Obstruction (range = 0 to 30) represents the extent to which various disruptions got in the way of valued living; higher scores represent more interference with living consistently with one's values. The baseline and day 90 VQ scores are reported.
Time Frame: Baseline, Day 90
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Change in Depression Score, as Measured by PHQ-9 Assessment
Description: The PHQ-9 consists of 9 items, each of which is scored 0 to 3, giving a 0 to 27 severity score
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Change in Cognitive Function, as Measured by PROMIS Cognitive Function Assessment
Description: as for outcome 15
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Change in Cognitive Function, as Measured by Montreal Cognitive Assessment
Description: This administered assessment is subdivided into visuospatial/executive (5pts), naming (3pts), memory (no points), attention(5pts), language(3pts), abstraction(2pts), delayed recall(5pts), and orientation(6pts). All the subdivided sections have as many questions as they have points. For analysis, the cut point is if the patient has less than 26 points.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Change in Physical Function, as Measured by PROMIS Physical Function Assessment
Description: as for outcome 15
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Change in Physical Function, as Measured by PROMIS Fatigue Assessment
Description: as for outcome 15
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

46. Other Pre Specified Outcome: Number of Falls, as Assessed by Falls Questionnaire
Description: Participants will answer Yes/No to whether they have had any falls in the preceding 6 months
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

47. Other Pre Specified Outcome: Change in Step Count, as Measured by Activity Tracker
Description: Activity tracker tracks number of steps per day
Time Frame: Continuous from baseline up to 3 years
Reporting Status: Not Posted

48. Other Pre Specified Outcome: Change in Physical Function, as Measured by 30 Second Sit-stand
Description: Subjects will sit in a chair with their arms crossed over their chest and rise to a standing position, then return to seated position. They will repeat this as many times as they can in 30 seconds.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

49. Other Pre Specified Outcome: Change in Physical Function, as Measured by Short Physical Performance Battery (SPPB)
Description: All the task points are added which make the SPPB score. The cut-point for the SPPB is a score of 10. The cumulative and sections scores are assessed individually and comprehensively. This assessment score will be used as a tool for evaluating lower extremity functioning in older persons.
Time Frame: Baseline, Day 30, Day 90, Day 180, Year 1, Year 2, and Year 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for participants continuously from enrollment through Year 3
Description: Adverse events are self-reported by study participants. The patients on this study are undergoing allogeneic stem cell transplantation, which is a procedure that is associated with high rates of adverse outcomes and morbidity. As such, we only record adverse events that are directly reported to us by the study participant or that are directly related to the study activity (i.e. falls during 6 minute walk test, emotional distress from answering study questionnaires, etc.)
Groups:
- Caregivers: 14 HCT patients caregivers at Duke
  Acceptance and Commitment Therapy (ACT): The ACT sessions will be tailored to the clinical challenges of HCT. Sessions are with a mental health professional and are 45-60 minutes in duration and include both the participant and caregiver.
Arm/Group | Hematopoietic Stem Cell Transplantation (HCT) Patients | Caregivers
All-Cause Mortality (participants affected / at risk) | 4/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT04423939/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT04423939/ICF_000.pdf